CLINICAL TRIAL: NCT03363022
Title: To Assess the Role of Fecal Microbiota Transplant in Acute Liver Failure- A Double Blind Controlled Trial
Brief Title: To Assess the Role of Fecal Microbiota Transplant in Acute Liver Failure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Funds
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-ALF-04
Record Dates: First submitted 2017-09-23; First posted 2017-12-05 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Acute Liver Failure
MeSH Terms: conditions — Liver Failure, Acute | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Medical Treatment+Fecal Microbiota Transplant (Experimental)
  Interventions: Drug: Standard Medical Treatment; Other: Fecal Microbiota Transplant
- Standard Medical Treatment+Placebo (Active Comparator)
  Interventions: Drug: Standard Medical Treatment; Other: Placebo

INTERVENTIONS:
Drug: Standard Medical Treatment — Standard Medical Treatment includes antibiotics,CRRT (Continuous Renal replacement Therapy),Liver Dialysis.
Other: Fecal Microbiota Transplant — Fecal Microbiota Transplant Stool specimen (preferably Bristol Stool Type 3 or 4) with a weight of ∼50 g will be considered adequate.
  250 mL sterile normal saline will be added to the stool sample and homogenized with a blender for 2-4minutes in pulses of 30 seconds with 10 seconds wait in between each pulse.
  Enema to be held for 30 minutes.
  Arms: Standard Medical Treatment+Fecal Microbiota Transplant
Other: Placebo — Placebo will be identical and non medicinal to the Fecal Microbiota Transplant
  Arms: Standard Medical Treatment+Placebo

SUMMARY:
All patients of Acute liver failure not meeting the KCH (King's College Hospital) criteria/or meeting KCH criteria not having option of liver transplant will be recruited for the trial. The first group will receive Standard medical care with Fecal Microbiota transplant on Day 1 for 3 consecutive days. FMT (Fecal Microbiota Transplant) will be delivered rectally which will be placed bedside. Suitable donor will be screened and the stool samples will be used as per criteria. Stool samples will be taken at the time at Day 0, 1(Post FMT), Day 4, 6, 14,21. Sepsis screen will be sent. Inflammatory markers will be sent on Day 0,1, 4,6, 14,21. The second group will receive standard medical therapy/and an placebo. Stool samples will be sent on Day 0,1, 4, 6 , 14,21. Inflammatory markers will be sent on the time on day 0,1 4,6 , 14,21.

ELIGIBILITY:
Inclusion Criteria:

Acute liver failure -Not meeting KCH Criteria/Meeting KCH Criteria but not having Liver transplant option

Exclusion Criteria:

1. Culture Positive Sepsis
2. History of taking lactulose, rifaximin, neomycin, metronidazole, L-Ornithine L-Aspartate
3. Receiving psychoactive drugs, promotility and hypomotility drugs
4. Pregnant females

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival in both groups | Day 21

SECONDARY OUTCOMES:
Resolution of SIRS (Systemic Inflammatory Response Syndrome) in both groups | Day 1,2,5,7,14,21
Reduction of ammonia in both groups | Day 1,2,5,7,14,21
Improvement of Cerebral edema in both groups | Day 1,2,5,7,14,21
  Improvement is defined as transcranial doppler < 0.9/Features suggestive of edema in CT imaging
Improvement in SOFA (Sequential Organ Failure Assessment) Score in both groups | Day 21

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No